CLINICAL TRIAL: NCT03901365
Title: The Effect of Neuroplastic Pain Education on Quality of Life in Patients with Chronic Low Back Pain Who Treated Via Manual Therapy: a Single Blind Randomized Controlled Study
Brief Title: The Effect of Neuroscience Pain Education on Quality of Life in Patients with Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principal Investigator,, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KutahyaMSUFTR
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low Back Pain; Quality of Life; Pain
Keywords: Manual Therapy; Neuroscience pain education; Quality of life; Chronic low back pain
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Patient received manual therapy in addition neuroscience pain education sessions
  Interventions: Other: Neuroscience pain education; Other: Manual therapy
- Group 2 (Active Comparator): Patient received manual therapy in addition tradition education sessions
  Interventions: Other: Traditional patient education; Other: Manual therapy

INTERVENTIONS:
Other: Neuroscience pain education — In Neuroscience pain education (NPE) sessions, patients were informed about the pain experience and the neurophysiological process about pain. NPE was performed by the method proposed by Louw et al (12). NPE was administered 4 sessions per week for four weeks. Trainings were conducted in the form of face-to-face interview and 45-50 minutes of one-to-one sessions.
  Arms: Group 1
Other: Traditional patient education — In traditional patient education (TPE) sessions were aimed to explain to patients a proposed treatment or efficacy of a certain manual therapy technique or approach, have focused heavily on biomechanical and anatomical models. These models would imply that injury, disease, and muscle guarding may lead to altered movement patterns, asymmetrical loading, and resultant pain and dysfunction. TPE was administered 4 sessions per week for four weeks. Trainings were conducted in the form of face-to-face interview and 45-50 minutes of one-to-one sessions.
  Arms: Group 2
Other: Manual therapy — Manual therapy (MT) was individualized according to each patient's response to treatment. In this method, the physiotherapist identifies and performs techniques suitable for the patient's symptoms. If the selected techniques do not have a direct positive effect on the patient's symptoms, they are replaced with other techniques.MT were performed in a total of 8 sessions, held twice a week for 4 weeks. Treatment sessions lasted an average of 40-45 minute.The entire treatment program was carried out by the same physiotherapist who is trained and experienced in this area.

SUMMARY:
Manual therapy are among the therapeutic approaches frequently used in chronic low back pain (CLBP). Although most clinicians conduct patient education according biomedical model of pain, a relatively new approach which is referred to as neuroscience pain education (NPE) is promising in patients with CLBP. Therefore the aim of this study was to investigate whether NPE in patients with CLBP who treated via manual therapy technique will produce different outcomes in terms of pain severity and QoL compared to traditional patient education.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study.
* Patients with 18-65 years
* Had low back pain for at least 6 months,
* Reported pain severity of 5 or greater according to the numeric pain rating scale

Exclusion Criteria:

* Previous spine or lower extremity surgery
* Severe osteoporosis
* Spondyloarthropathy
* Spondylolisthesis
* Lumbar stenosis
* Lumbar fractures
* Malign tumor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL): Turkish Short form-36 (SF-36) questionnaire | Change from Baseline SF-36 at 4th weeks.
  All patients additionally completed Turkish Short form-36 (SF-36) questionnaire, 36-item generic self-administered instrument that consists of eight subscales relating to various aspects of the QoL: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health. The eight subscales are scored from 0 to 100, with higher scores indicating better health status

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Change from Baseline NPRS at 4th weeks.
  The NPRS was used to assess the participants' pain levels. In the NPRS, patients are asked to verbally rate the severity of their pain on a scale from 0 to 10. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme.

CONTACTS AND LOCATIONS:
Locations (1):
- Yoncali Physical Therapy and Rehabilitation Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No